CLINICAL TRIAL: NCT00303849
Title: Phase I/II Study of Carboplatin, Melphalan and Etoposide Phosphate in Conjunction With Osmotic Opening of the Blood-Brain Barrier and Delayed Intravenous Sodium Thiosulfate Chemoprotection, in Previously Treated Subjects With Anaplastic Oligodendroglioma or Oligoastrocytoma
Brief Title: Carboplatin, Melphalan, Etoposide Phosphate, Mannitol, and Sodium Thiosulfate in Treating Patients With Previously Treated Brain Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00002868; NCI-2013-00786 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CR00002456; 2868; IRB00002868 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Anaplastic Oligoastrocytoma; Anaplastic Oligodendroglioma; Mixed Glioma; Oligoastrocytoma
MeSH Terms: conditions — Oligodendroglioma; Glioma; Astrocytoma | interventions — Carboplatin; Etoposide; etoposide phosphate; Mannitol; Melphalan; sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (etoposide, mannitol, melphalan, carboplatin, STS) (Experimental): Patients receive etoposide phosphate IV over 10 minutes, mannitol IA over 30 seconds, melphalan IA over 10 minutes, and carboplatin IA over 10 minutes on days 1 and 2. Patients then receive sodium thiosulfate IV over 15 minutes at 4 and 8 hours after carboplatin. Courses repeat every 4 to 6 weeks for up to 12 months.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Etoposide Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mannitol; Drug: Melphalan; Other: Quality-of-Life Assessment; Drug: Sodium Thiosulfate

INTERVENTIONS:
Drug: Carboplatin — Given IA
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mannitol — Given IA
  Other Names: D-Mannitol; Mannitol, D-; Osmitrol; Resectisol
Drug: Melphalan — Given IA
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Sodium Thiosulfate — Given IV
  Other Names: Cyanide Antidote Package; Disodium Thiosulfate; S-Hydril; Sodium Hyposulfate; Sodium Thiosulfate Pentahydrate; Sodium Thiosulphate; Sodothiol; Thiosulfate, Sodium, Pentahydrate; Thiosulfuric acid disodium salt

SUMMARY:
This phase I/II trial studies the side effects and best dose of melphalan when given together with carboplatin, etoposide phosphate, mannitol, and sodium thiosulfate and to see how well they work in treating patients with previously treated brain tumors. Drugs used in chemotherapy, such as melphalan, carboplatin, and etoposide phosphate, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing, or by stopping them from spreading. Osmotic blood-brain barrier disruption (BBBD) uses mannitol to open the blood vessels around the brain and allow cancer-killing substances to be carried directly to the brain. Sodium thiosulfate may help lessen or prevent hearing loss and toxicities in patients undergoing chemotherapy with carboplatin and BBBD. Giving carboplatin, melphalan, etoposide phosphate, mannitol, and sodium thiosulfate together may be an effective treatment for brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate toxicity and estimate the maximum tolerated dose (MTD) of melphalan (intra-arterially [i.a.]) administered in conjunction with carboplatin (i.a.) and etoposide phosphate (intravenously [i.v.]) undergoing BBBD, in subjects with anaplastic oligodendroglioma or oligoastrocytoma. (Phase I) II. To examine the efficacy (one year progression free survival [1YPFS]) of carboplatin (i.a.), melphalan (i.a.) and etoposide phosphate (i.v.) in conjunction with BBBD, in subjects with anaplastic oligodendroglioma or oligoastrocytoma. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the incidence of severe neutropenia (specifically febrile neutropenia or sepsis) of carboplatin (i.a.), melphalan (i.a.) and etoposide phosphate (i.v.) in conjunction with BBBD, in subjects with anaplastic oligodendroglioma or oligoastrocytoma.

II. To evaluate the overall toxicity of carboplatin (i.a.), melphalan (i.a.), and etoposide phosphate (i.v.) in conjunction with BBBD.

III. To estimate the differences in tumor response, 1YPFS and survival, in subjects with allelic loss of chromosomes 1p and 19q, and tumor protein p53 (p53) immunocytochemistry, versus subjects without allelic loss.

IV. To assess quality of life, cognitive function, and performance status of subjects undergoing treatment with carboplatin, melphalan and etoposide phosphate in conjunction with BBBD.

V. To estimate differences in 1YPFS between subjects with anaplastic oligodendroglioma and patients with oligoastrocytoma.

VI. To describe the role of biopsy versus extent of surgery (sub-maximal versus maximal safe resection) on 1YPFS and survival.

VII. To describe the role of prior radiation on tumor response, 1YPFS and survival.

OUTLINE: This is a phase I, dose-escalation study of melphalan followed by a phase II study.

Patients receive etoposide phosphate IV over 10 minutes, mannitol IA over 30 seconds, melphalan IA over 10 minutes, and carboplatin IA over 10 minutes on days 1 and 2. Patients then receive sodium thiosulfate IV over 15 minutes at 4 and 8 hours after carboplatin. Courses repeat every 4 to 6 weeks for up to 12 months.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with pathologic evidence of an anaplastic oligodendroglioma or mixed glioma (i.e. oligoastrocytoma) are eligible; histopathologic diagnosis will be made using World Health Organization classification criteria; to qualify as a mixed tumor there must be a minimum of 25% oligodendroglial element
* Surgical procedure may have been complete resection, partial resection, or biopsy
* Subjects must have had prior treatment with temozolomide; at least 28 days must have elapsed since completion of temozolomide or other chemotherapy
* If subject has not undergone radiation therapy, then subject must have undergone prior consultation with a radiation oncologist (who is not an investigator on this study); if the subject has undergone radiation therapy, then at least 14 days must have elapsed since completion of radiation
* Subjects performance status must be (Karnofsky performance status [KPS] greater than or equal to 50; Eastern Cooperative Oncology Group [ECOG] less than or equal to 2)
* White blood cell count >= 2.5 x 10^3/mm^3
* Absolute granulocyte count > 1.5 x 10^3/mm^3
* Platelets >= 100 x 10^3/mm^3
* Serum creatinine < 1.5 x upper limit of normal
* Bilirubin < 1.5 x upper limit of normal
* Subjects baseline serum glutamic oxaloacetic transaminase (SGOT)/serum glutamate pyruvate transaminase (SGPT) must be < 2.5 x institutional upper limit of normal
* Subjects must sign a written informed consent in accordance with institutional guidelines
* The effects of carboplatin, melphalan and etoposide phosphate on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because these agents as well as other therapeutic agents used in this trial are known to be teratogenic. Sexually active women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study treatment and for the duration of study treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Subjects with radiographic signs of excessive intracranial mass effect with associated rapid neurologic deterioration, and/or spinal cord block
* Subjects at significant risk for general anesthesia
* Subjects with uncontrolled (over the last 30 days) clinically significant confounding medical conditions
* Subject is pregnant, has a positive serum human chorionic gonadotropin (hCG) or is lactating
* Subjects who have contraindications to carboplatin, melphalan, etoposide phosphate, or sodium thiosulfate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-09-15 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
MTD of melphalan, defined as one dose level below the dose that produces grade 4 toxicity in 33% of patients, graded in accordance with National Cancer Institute Common Toxicity Criteria (NCI CTC) (version 3.0) (Phase I) | 4 weeks
Overall survival | 1 year
Progression free survival (Phase II) | 1 year
  Kaplan-Meier method will be used. 95% confidence intervals estimated. Cox proportional hazards regression models will be fit to explore potential predictors.
Response rate | 1 year
Time to best response | 1 year

SECONDARY OUTCOMES:
Functional outcomes | 1 year
  Descriptive numeric and graphical summaries for functional status, quality of life, and cognitive function will be estimated for all subjects and separately for subjects with anaplastic oligodendrogliomas and oligoastrocytomas.
Incidence of severe neutropenia (specifically febrile neutropenia or sepsis) in accordance with NCI CTC (version 3.0) | 1 year
  Incidence rates of grade III/IV events and associated 95% confidence intervals will be estimated.
Rates of two year progression free survival (2YPFS) for specific tumor types | 2 years
  Separate estimates of 2YPFS and overall survival (and associated confidence intervals) will be made for subjects with anaplastic oligodendroglioma and for subjects with oligoastrocytoma. Confidence intervals will also be used to describe differences between this subject series and our earlier subject series.

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Neuwelt, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - OHSU Knight Cancer Institute, Portland, Oregon